CLINICAL TRIAL: NCT04634630
Title: The Influence of Cancer Stem-cells on Risk of Relapse in Patients Harboring Adenocarcinoma and Squamous Cell Carcinoma of the Lung: a Prospective Cohort Study
Brief Title: The Influence of Cancer Stem-cells on Risk of Relapse in Patients Harboring Adenocarcinoma and Squamous Cell Carcinoma of the Lung
Status: Completed | Type: Observational
Sponsor: Beatrice Aramini (Other)
Responsible Party: Sponsor-Investigator, Beatrice Aramini, Assistant Professor in Thoracic Surgery, Azienda Ospedaliero-Universitaria di Modena
Organization: Azienda Ospedaliero-Universitaria di Modena (Other)
Other Study IDs: STEMCELL/1
Record Dates: First submitted 2020-11-12; First posted 2020-11-18 (Actual); Last update posted 2021-06-01 (Actual); Status verified 2021-05

CONDITIONS: Lung Cancer, Nonsmall Cell; Relapse/Recurrence; CSC
Keywords: Non Small Cell Lung Cancer; Cancer Stem Cells
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Genetic: Exposure to lung cancer stem cells — The exposure to lung cancer stem cells was measure as the percentage of Aldehyde dehydrogenase (ALDH) on all viable cells extracted from surgically resected tumor specimens

SUMMARY:
The present study is a prospective cohort study. The aim is to assess the relationship between the presence of cancer stem-cells (CSC) and the risk of relapse in patients with early and locally advanced adenocarcinoma and squamous cell carcinoma of the lung

ELIGIBILITY:
Inclusion Criteria:

* patients with stage I, II or IIIA adenocarcinoma of squamous cell carcinoma of the lung
* age between 18 and 85
* R0 resection
* availability of formalin-fixed, paraffin-embedded surgery specimen from the primary tumor
* availability of fresh surgical specimen for cytofluorimetric analysis

Exclusion Criteria:

* incomplete resection
* unknown tumor, node or metastasis status
* synchronous tumors
* previous lung cancer

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent major lung resection by lateral thoracotomy or videothoracoscopic approach for stage I, II, or IIIA adenocarcinoma or squamous cell carcinoma of the lung (tumor, node, metastasis (TNM) staging system, eighth edition)
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2017-10-17 (Actual); Primary Completion 2020-10-17 (Actual); Study Completion 2020-10-17 (Actual)

PRIMARY OUTCOMES:
Relapse Free Survival | Minimum follow-up time: 1 year
  Days from lung cancer resection to relapse

CONTACTS AND LOCATIONS:
Overall Officials: Uliano Morandi, MD, Principal Investigator — Azienda Ospedaliero-Universitaria di Modena
Locations (1):
- Azienda Ospedaliero-Universitaria di Modena, Modena, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Masciale V, Banchelli F, Grisendi G, D'Amico R, Maiorana A, Stefani A, Morandi U, Stella F, Dominici M, Aramini B. Cancer Stem Cells and Cell Cycle Genes as Independent Predictors of Relapse in Non-small Cell Lung Cancer: Secondary Analysis of a Prospective Study. Stem Cells Transl Med. 2022 Aug 23;11(8):797-804. doi: 10.1093/stcltm/szac040. PMID 35674389
- [Derived] Masciale V, Banchelli F, Grisendi G, D'Amico R, Maiorana A, Stefani A, Morandi U, Stella F, Dominici M, Aramini B. The Influence of Cancer Stem Cells on the Risk of Relapse in Adenocarcinoma and Squamous Cell Carcinoma of the Lung: A Prospective Cohort Study. Stem Cells Transl Med. 2022 Mar 31;11(3):239-247. doi: 10.1093/stcltm/szab029. PMID 35356974